CLINICAL TRIAL: NCT06325137
Title: Transcriptome Analysis in Idiopathic Nephrotic Syndrome: an Insight Into the Mechanisms of Steroid Responsiveness
Brief Title: Transcriptome Analysis in Idiopathic Nephrotic Syndrome: Steroid Responsiveness
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 24/2022
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Nephrotic Syndrome
Keywords: Whole transcriptome sequencing; Idiopathic nephrotic syndrome pathogenesis; Steroid responsiveness prediction
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Transcriptome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with steroid-resistant nephrotic syndrome: Identification of a possible molecular signatures at t0 by whole transcriptome analysis from PBMCs
  Interventions: Diagnostic Test: Transcriptome analyses
- Patients with steroid sensitive nephrotic syndrome: Identification of a possible molecular signatures at t0 by whole transcriptome analysis from PBMCs
  Interventions: Diagnostic Test: Transcriptome analyses

INTERVENTIONS:
Diagnostic Test: Transcriptome analyses — A sample of peripheral whole blood cells will be collected at the onset before the initiation of steroid treatment (time 0, t0) and after 6 weeks at the definition of steroid sensitivity/unresponsiveness (time 1, t1).

SUMMARY:
Idiopathic nephrotic syndrome (INS) affects the glomerular barrier by damaging the podocytes with foot process effacement, leading to a pathological increase of permeability and protein loss. INS classification is based on the clinical response to glucocorticoid (GC) therapy. When GCs treatment fails to induce remission in a four-six weeks course, patients are defined as affected with steroid-resistant nephrotic syndrome (SRNS).

The whole transcriptome sequencing could consent the INS classification at onset, prior to glucocorticoids (GCs) treatment, allowing to reduction of unuseful GCs treatment. RNA sequencing technologies allow an extensive characterization of the transcriptomic profile and permit global changes in gene expression levels between different conditions such as active and remission of the disease.

Of great interest is the research of a molecular biomarker to predict steroid resistance, a predictor that is not yet available. Among the candidate biomarkers, pharmacogenomic determinants are promising, even if available studies are still limited. Among these, some epigenetic factors have been previously suggested. Data obtained in animal models suggests that nucleotide-binding oligomerization domain-like receptors (NOD-like receptor) pyrin domain containing 3 (NLRP3) inflammasome can be deregulated in a wide variety of glomerular diseases, including those causing INS. Another potential marker involved in steroid response is the long noncoding RNA GAS5. Data reported in the literature indicate that abnormal levels of GAS5 in peripheral blood mononuclear cells (PBMCs) may alter steroid effectiveness in autoimmune diseases, such as inflammatory bowel disease.

Preliminary findings show that the study of NLRP3 promoter methylation could be reduced in the blood of SRNS compared with steroid-sensitive nephrotic syndrome (SSNS) patients. Moreover, unpublished encouraging results on the association between Growth Arrest Specific 5 (GAS5) expression and steroid response in INS in PBMCs were obtained in a preliminary study conducted on 8 patients with the first episode of INS. PBMCs were obtained and GAS5 gene expression was evaluated using TaqMan technology. Patients affected with SRNS presented significantly higher levels of GAS5 in comparison with the SSNS group. In PBMCs from SRNS patients, the GAS5 expression could reduce the availability for binding to GCs target genes of the activated GCs receptor and suppresses GC transcriptional activity.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of INS
* age 1 - 12 years
* signed informed consent by parents or legal guardians
* For controls: aged-matched individuals with Congenital Anomalies of the Kidney and Urinary Tract (CAKUT)

Exclusion Criteria:

* Patients aged <1 year or > 12 years
* Patients diagnosed with a secondary or genetic form of NS
* For controls: the presence of coexisting chronic kidney failure, autoimmune or autoinflammatory disease, or endocrinologic disorders.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with nephrosic syndrome
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Between groups differences in molecular signature by whole transcriptome analysis | At enrolment (T0)
  A sample of peripheral whole blood cells will be collected at the onset before the initiation of steroid treatment (time 0, t0)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided